CLINICAL TRIAL: NCT03221803
Title: Patient Satisfaction and Bone Changes in Bilateral Distal Extension Case Using OT Cap Versus OT Vertical Attachment "Randomized Clinical Trial"
Brief Title: Patient Satisfaction and Bone Changes for OT Cap and OT Vertical Attachment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ali Hassaan, Assistant lecturer at faculty of dentistry fayoum university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OT Cap_OT Vertical
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Patient Satisfaction; Bone Changes
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OT Vertical attachment (Experimental): The attachment consists of a male part that is in the form of a steady with a central hole. This part is attached to the abutments .the female component is a white standard retentive clip engaging the outer walls of a steady male. It is incorporated in the partial denture together with a castable balancing pin that fits into the central hole of the steady male and aids in centering the prosthesis during the final stage of insertion; thereby ensuring a longer life to the retentive clips.
  Interventions: Other: OT Vertical attachment
- OT Cap attachment (Active Comparator): Beveled castable bar with micro-size sphere located in first molar region, and attached to the distal surface of the waxed crowns to be cast as one piece, Nylone caps of standard retention for micro size sphere this nylon caps fit onto their spheres and located in metal housing at fitting surface on the denture and Positioning rings to maintain the space for nylon cap during construction of the partial denture metal framework.
  Interventions: Other: OT cap attachment

INTERVENTIONS:
Other: OT Vertical attachment — new extra coronal castable attachment
  Other Names: Castable twin cylinder attachment
  Arms: OT Vertical attachment
Other: OT cap attachment — standard extra coronal attachment
  Other Names: extra coronal castable attachment
  Arms: OT Cap attachment

SUMMARY:
The purpose of this study aimed to answer a clinical question whether In a patient with bilateral distal extension area, would the metal framework partial denture with OT vertical attachment versus partial denture with OT CAP attachment result in better patient satisfaction?

ELIGIBILITY:
Inclusion Criteria:

* patients age ranged between 35-45years old.
* All patients have Kennedy class I partially edentulous mandibular arch in which the last remaining teeth were the second premolars bilaterally.
* The abutment teeth had an apparently good periodontal condition with no signs of mobility or inflammation with firm and healthy mucosa.
* Edentulous ridge covered by health firm mucoperiosteum, without abnormal bony irregularity or severe lingual undercuts.
* Patients with normal relationship of maxilla and mandible (Angle class I ridge classification) and sufficient inter-arch space (6mm) the size of the attachment
* The opposing dentition is intact arch with no noticeable over eruption or tilting or restored with acceptable fixed restoration.
* All patients are free from neurological, muscular disorders and tempro-mandibular joint disorders.
* Only patients who can be easily motivated to achieve and maintain good oral

Exclusion Criteria:

* Patient with limited skills
* Un co-operative patients.
* patient with bad oral hygiene

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction assessed using questionnaire | 9 months
  Questionnaire for patient satisfaction

SECONDARY OUTCOMES:
bone height | 9 months
  radio graphically by digora
bone density | 9 months
  radio graphically by digora

IPD SHARING:
Plan to Share IPD: Undecided